CLINICAL TRIAL: NCT05086224
Title: Hematoma Block vs. Bier Block: Which is More Effective for Closed Fracture Reduction?
Brief Title: Hematoma Block Versus Bier Block for Closed Fracture Reduction
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lucas Marchand, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 131997
Record Dates: First submitted 2021-09-16; First posted 2021-10-20 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Distal Radius Fractures
Keywords: Distal radius fractures; Hematoma block; Bier block; Pain
MeSH Terms: conditions — Wrist Fractures; Pain | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hematoma Block (Other): Inject 20 mL of 1% lidocaine without epinephrine into the hematoma site.
  Interventions: Drug: Hematoma Local Anesthetic Block Procedure with 1% Lidocaine
- Bier Block (Other): Intravenous administration a maximum lidocaine dose of 3 mg/kg.
  Interventions: Drug: Bier Anesthetic Block Procedure with 1% Lidocaine

INTERVENTIONS:
Drug: Hematoma Local Anesthetic Block Procedure with 1% Lidocaine — Inject anesthetic into the hematoma site, 20 mL of 1% lidocaine without epinephrine.
  Other Names: Lignocaine, Xylocaine, Ztlido (lidocaine)
  Arms: Hematoma Block
Drug: Bier Anesthetic Block Procedure with 1% Lidocaine — Intravenous anesthetic infusion, a maximum lidocaine dosing of 3 mg/kg.
  Other Names: Lignocaine, Xylocaine, Ztlido (lidocaine)
  Arms: Bier Block

SUMMARY:
The investigators objective of this study is to evaluate the effectiveness of hematoma block versus intravenous regional anesthesia (Bier block) during closed reduction of distal radius fractures.

DETAILED DESCRIPTION:
The investigators objective of this study is to evaluate the effectiveness of hematoma block compared to intravenous regional anesthesia (Bier block) during closed reduction of distal radius fractures. Distal radius fractures represent one of the most commonly treated skeletal injuries in the US. Achieving a fracture reduction that restores anatomy of the distal radius is of paramount importance. Reductions that re-establish anatomical parameters can prevent a patient from requiring operative intervention for the fracture, eliminating the risks as well as costs that are inherent in undergoing surgery.

Intravenous regional anesthesia (IVRA) or 'Bier block' is an effective technique used to provide anesthesia to the distal extremity. IVRA involves venous infiltration of a local anesthetic with concomitant use of a tourniquet to restrict infiltration solely to the intended extremity. Hematoma block involves local infiltration of local anesthetic directly into the site of a hematoma to provide analgesia. Both IVRA and hematoma blocks can be used to provide analgesia during a variety of procedures including fracture manipulation and reduction, but there is a paucity of data regarding the possible superiority of one means of analgesia.

To date, only a few comparative studies has been performed regarding the use of these two analgesia methods. Numerous investigators have conducted studies evaluating these two methods of analgesia; but these studies were of relatively poor quality, are older (prior to 1995) or did not individually look at all radiographic parameters that are important to orthopedic surgical providers when determining if a distal radius fracture needs surgery, particularly ulnar variance and articular step-off or gapping.

The investigators institution is one of the few in the country that utilizes bier blocks, performed by orthopedic residents, for most closed reductions in the emergency department. This quality makes the investigators institution uniquely qualified and motivated to perform the proposed investigation.

Concerns regarding the implementation of the Bier block surround its' safety profile, including possible increased risk of carpal tunnel, and in more severe cases, seizures or cardiac arrest. Despite the frequency with which investigators manage distal radius fractures, our experience has been that the major complication profile of this technique is minimal. Other studies have supported the notion that catastrophic complications are rare and the most common "complication" is tourniquet pain. These studies are limited by their nature in that anesthesia or emergency medicine providers performed the Bier blocks, while in most instances having the orthopaedic provider perform the block as well as the reduction is more efficient.

The standard of care for most institutions is to perform a closed reduction of distal radius fracture with general conscious sedation or a local hematoma block. The investigators standard of care is to perform Bier blocks as the investigators believe it results in a more anatomic reduction, due to better analgesia and patient comfort during the procedure, thus allowing for more aggressive yet tolerable manipulation. Improved reduction quality may result in less conversion from closed management in a cast to surgical intervention which has direct impact on the patients being treated as well as on the health care system at large. The investigators hypothesis is that there is both better analgesia and fracture reduction with use of Bier block compared to hematoma block.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18+ years of age) with a closed distal radius.
* Eligible patients will be those who require a closed reduction for a displaced fracture.
* Any distal radius that falls outside of normal anatomic parameters will require reduction.
* Normal anatomic parameters include radial inclination: 22°; mean, 19° to 29°, radial height: 11 to 12 mm, and volar tilt 11°; mean,11° to 14.5°.
* Patients presenting with intact neurovascular exam will be included (sensation intact about ulnar, median, and radial nerve distributions with an intact radial pulse.

Exclusion Criteria:

* Not able to provide informed consent (intubated or cognitively impaired).
* Member of vulnerable populations such as non-English speaking and incarcerated patients.
* Pregnant or lactating women.
* Have open fractures or altered neurovascular exams.
* Have any confounding injures such as an associated dislocation or subluxation of the carpus or patients who have a concomitant upper extremity injury requiring surgery.
* Patients who will obtain follow-up elsewhere (as they will not be able to be studied longitudinally.
* Patients who have are unable to tolerate the tourniquet pressure while awake or in whom IV access is unable to be obtained in the correct hand will be excluded from the bier block arm of the study.
* Patients with skin compromise or breakdown or active infection overlying fracture site will be excluded from the hematoma block arm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) pain | Prior to fracture manipulation
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | During anesthetic injection or infusion, an average of 10 minutes.
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | During fracture manipulation, an average of 10 minutes.
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 30 minutes following fracture manipulation
  VAS pain score (0 no pain - 10 severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Marchand, MD, Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States